CLINICAL TRIAL: NCT01534195
Title: A Phase 4, Randomized, Double-Masked, Single Center, Placebo-Controlled Adaptive Clinical Trial, Using Prednisolone Sodium Phosphate Ophthalmic Solution, 1%, in Subjects With Allergic Conjunctivitis to Evaluate a Modified Conjunctival Allergen Challenge (CAC) Model
Brief Title: Evaluation of the Efficacy of Topical Ophthalmic Steroids in a Modified Conjunctival Allergen Challenge (CAC) Model
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ORA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 12-270-0001
Record Dates: First submitted 2012-01-25; First posted 2012-02-16 (Estimated); Results first posted 2019-01-15 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2012-07

CONDITIONS: Allergic Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prednisolone (Experimental): Prednisolone Sodium Phosphate Ophthalmic Solution, 1%
  Interventions: Drug: Prednisolone Sodium Phosphate Ophthalmic Solution 1%
- Placebo (Placebo Comparator): Tears Naturale II Ophthalmic Solution, 1%
  Interventions: Drug: Tears Naturale II Ophthalmic Solution

INTERVENTIONS:
Drug: Prednisolone Sodium Phosphate Ophthalmic Solution 1% — One drop in each eye, four times/day for 8 days.
  Arms: Prednisolone
Drug: Tears Naturale II Ophthalmic Solution — one drop in each eye, four times/ day (QID) for 8 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effectiveness of the modified Conjunctival Allergen Challenge (CAC) and observe how the produced allergic inflammation reacts to treatment with a proven ocular anti-inflammatory medication,

Prednisolone, assessed by the following measures:

* Ocular itching
* Conjunctival redness

DETAILED DESCRIPTION:
Prospective, single center, randomized, double-masked, placebo controlled study. Subjects will be randomized to one of the following treatment arms to dose four times per day (QID) for 8 days between Visits 4 and 5.

* Prednisolone phosphate
* Tears Naturale II Ophthalmic Solution (Placebo)

Duration:

Approximately 19 days

Controls:

Artificial Tears (Tears Naturale® II)

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age & either sex, any race
* Willing and able to follow all instructions
* Positive history of ocular allergies
* Reproducible positive ocular allergic reaction induced by conjunctival allergen challenge

Exclusion Criteria:

* Have planned surgery during trial period
* Female currently pregnant, planning a pregnancy or lactating
* Use of disallowed medications
* Have ocular infections, or ocular conditions that could affect study parameters
* Have moderate to severe dry eye
* Have used an investigational drug or device within 30 days of start of study
* Female that is currently pregnant, planning a pregnancy or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-01; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Shazly, MD, Principal Investigator — Ophthalmic society of Egypt, Egyptian Glaucoma Society, American Acadamy of Ophthalmology, American Glaucoma Society, The association for research in vision and ophthalmology, international society of refractive surgery, Pan Arab Glaucoma Society
Locations (1):
- Andover Eye Associates, Andover, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Prednisolone: Prednisolone Sodium Phosphate Ophthalmic Solution, 1%
  Prednisolone Sodium Phosphate Ophthalmic Solution 1%: One drop in each eye four times/day (QID) for 8 days.
- Placebo: Tears Naturale II Ophthalmic Solution, 1%
  Tears Naturale II Ophthalmic Solution: one drop in each eye QID for 8 days
Period: Overall Study
Arm/Group | Prednisolone | Placebo
Started | 5 | 6
Completed | 4 | 5
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Prednisolone: Prednisolone Sodium Phosphate Ophthalmic Solution, 1%
  Prednisolone Sodium Phosphate Ophthalmic Solution 1%: One drop in each eye QID for 8 days.
- Total: Total of all reporting groups
Arm/Group | Prednisolone | Placebo | Total
Number analyzed (Participants) | 4 | 5 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 8
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.6 (6.693) | 49.5 (13.329) | 49.55 (8.896)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Ocular Itching Change From Baseline to Day 11
Description: Ocular itching, as assessed by the participant, was measured on a 4-point scale 5 minutes after the conjunctival allergen challenge (CAC). 0 was best (no itching), and 4 was worst (worst itching).
Time Frame: 5 minutes post-CAC
Population: All participants who completed the study
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prednisolone | Placebo
Number analyzed (Participants) | 4 | 5
units on a scale | -1.1 (0.14) | -0.45 (0.86)

2. Secondary Outcome: Conjunctival Redness Change From Baseline to Day 11
Description: Conjunctival Redness, as measured by the investigator, on a 4-point scale 7 minutes after the CAC. 0 was best (no redness), and 4 was worst (most redness)
Time Frame: 7 Minutes post-CAC
Population: All participants who completed the study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prednisolone | Placebo
Number analyzed (Participants) | 4 | 5
score on a scale | -0.69 (0.31) | 0.40 (0.88)

3. Secondary Outcome: Episcleral Redness Change From Baseline to Day 6
Description: Episcleral redness, as measured by the investigator, on a 4-point scale 7 minutes after the CAC.0 was best (least redness), and 4 was worst (most redness).
Time Frame: 7 minutes post-CAC
Population: All participants who completed the study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prednisolone | Placebo
Number analyzed (Participants) | 4 | 5
score on a scale | -1.0 (0.41) | 0.45 (0.93)

4. Secondary Outcome: Ciliary Redness Change From Baseline to Day 6
Description: Ciliary redness, as measured by the investigator, on a 4-point scale 7 minutes after the CAC. 0 was best (least redness), and 4 was worst (most redness).
Time Frame: 7 minutes post-CAC
Population: All participants who completed the study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prednisolone | Placebo
Number analyzed (Participants) | 4 | 5
score on a scale | -0.94 (0.66) | 0.30 (0.96)

ADVERSE EVENTS:
Time Frame: AEs were collected from the date of informed consent to the date of the final visit (1 month).
Arm/Group | Prednisolone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/6
Other Adverse Events (participants affected / at risk) | 1/5 | 3/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prednisolone (N=5) | Placebo (N=6)
Mucous Discharge (OU) (Eye disorders) | 0 (0) | 2 (2)
Headache (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Backache (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No